CLINICAL TRIAL: NCT01832506
Title: A Japanese Multicenter, Open Label, Phase I Trial of c-Met Inhibitor MSC2156119J Given Orally as Monotherapy to Subjects With Solid Tumors
Brief Title: A Japanese Phase 1 Trial of c-Met Inhibitor MSC2156119J in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200095-003
Record Dates: First submitted 2013-04-05; First posted 2013-04-16 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; MSC2156119J; c-Met inhibitor; Japanese; Phase 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MSC2156119J (Experimental)
  Interventions: Drug: MSC2156119J

INTERVENTIONS:
Drug: MSC2156119J — Subjects will be administered with MSC2156119J 215 mg, 300 mg and 500 mg orally once daily for repeated 21-day cycles until disease progression or unacceptable toxicity.

SUMMARY:
This is a Japanese multicenter, open-label, Phase 1 study to evaluate safety and efficacy of MSC2156119J in subjects with malignant solid tumor which is refractory to standard therapy or to which no effective standard therapy is applicable.

ELIGIBILITY:
Inclusion Criteria:

* A subject with a histologically or cytologically confirmed diagnosis of malignant solid tumor which is refractory to standard therapy or to which no effective standard therapy is applicable
* An archived tumor tissue is available or biopsy of tumor tissues can be newly performed
* A Japanese male or female, age greater than or equal to (>=) 20 years
* A subject who has read the Subject Information Sheet and understood the details of this clinical trial, and is willing and able to give his/her informed consent.
* A female of child-bearing potential must have a negative blood pregnancy test result at her screening period. A female subject of child-bearing potential must be willing to avoid pregnancy by using an adequate method of contraception Life expectancy is at least 3 months
* Other inclusion criteria apply

Exclusion Criteria:

* Known Human immunodeficiency virus (HIV) positivity, active hepatitis C, or active hepatitis B
* Presence of liver fibrosis or liver cirrhosis that has been histologically diagnosed
* Signs or symptoms that suggest transmissible spongiform encephalopathy
* Received major surgery within 6 weeks before Day 1 in Cycle 1
* Known drug abuse or alcohol abuse
* Known hypersensitivity to any of the trial treatment ingredients
* Hematological test abnormalities
* Renal impairment as defined in the protocol
* Liver dysfunction as defined in the protocol
* History or presence of central nervous system metastasis
* History or presence of disease or condition that may hamper compliance or absorption of the investigational medicinal product (IMP) due to difficulty in swallowing or absorption
* Poor performance status of Eastern Cooperative Oncology Group Performance status (ECOG PS) >= 2
* Received any anti-cancer therapy days Received extensive prior radiotherapy that irradiates more than 30 percent of bone marrow
* Received any radiotherapy within 4 weeks before Day 1 in Cycle 1
* Pregnancy and lactation period
* History of receiving treatment with any c-Met signaling pathway inhibitor
* Participation in another interventional clinical trial within the past 30 days from Day 1 in Cycle 1
* Other significant disease that in the Investigator's opinion would exclude the subject from the trial
* Legal incapacity or limited legal capacity
* Other exclusion criteria apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., Japan
Locations (2):
- Japan (2):
  - Research site, Kashiwa
  - Research site, Shizuoka

REFERENCES:
- [Result] Shitara K, Yamazaki K, Tsushima T, Naito T, Matsubara N, Watanabe M, Sarholz B, Johne A, Doi T. Phase I trial of the MET inhibitor tepotinib in Japanese patients with solid tumors. Jpn J Clin Oncol. 2020 Aug 4;50(8):859-866. doi: 10.1093/jjco/hyaa042. PMID 32328660
- [Derived] Xiong W, Hietala SF, Nyberg J, Papasouliotis O, Johne A, Berghoff K, Goteti K, Dong J, Girard P, Venkatakrishnan K, Strotmann R. Exposure-response analyses for the MET inhibitor tepotinib including patients in the pivotal VISION trial: support for dosage recommendations. Cancer Chemother Pharmacol. 2022 Jul;90(1):53-69. doi: 10.1007/s00280-022-04441-3. Epub 2022 Jun 30. PMID 35771259
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=EMR%20200095-003
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): 15 April 2013/20 September 2013. Last subject completed: 22 October 2014.
Groups:
- MSC2156119J 215 mg: Subjects were administered with MSC2156119J 215 milligram (mg) orally once daily for repeated 21-day cycles until disease progression or unacceptable toxicity.
- MSC2156119J 300 mg: Subjects were administered with MSC2156119J 300 mg orally once daily for repeated 21-day cycles until disease progression or unacceptable toxicity.
- MSC2156119J 500 mg: Subjects were administered with MSC2156119J 500 mg orally once daily for repeated 21-day cycles until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Started | 3 | 3 | 6
Completed | 3 | 3 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects who had received at least 1 dose of the investigational medicinal product (IMP).
Groups:
- MSC2156119J 215 mg: Subjects were administered with MSC2156119J 215 mg orally once daily for repeated 21-day cycles until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg | Total
Number analyzed (Participants) | 3 | 3 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.6) | 62.0 (5.0) | 65.7 (9.8) | 63.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 2 | 2 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Dose Limiting Toxicity (DLT)
Description: DLT: defined using National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.0, as any of following toxicities: Grade 4 neutropenia for more than 7 days; greater than or equal to (>=) Grade 3 febrile neutropenia; Grade 4 or Grade 3 thrombocytopenia with bleeding; >=Grade 3 nausea despite adequate treatment; >=Grade 3 any non-hematological AE (DLT defined specifically for following cases: >=Grade 3 liver adverse event [AE] requiring recovery period of more than 7 days or to Grade 1 without liver metastases or Grade 2 with liver metastases ; >=Grade 3 lipase and/or amylase elevation with confirmation of pancreatitis. An isolated lipase and/or amylase elevation of >=Grade 3 without clinical/radiological evidence of pancreatitis was not classified as DLT); and >=Grade 2 any AE not otherwise defined as DLT that, due to prolonged recovery to Grade 1 (or less) or baseline status, led to delay of treatment with IMP for more than 21 days.
Time Frame: Cycle 1 (Day 1 up to 21)
Population: DLT analysis set included all subjects who completed Cycle 1 (having received 80% or more of planned cumulative dose of IMP for Cycle 1) or who stopped treatment with IMP during Cycle 1 because of DLT.
Measure: Number; unit: subjects
Groups:
- MSC2156119J 215 mg: Subjects were administered with MSC2156119J 215 mg once daily for repeated 21-day cycles until disease progression or unacceptable toxicity.
- MSC2156119J 300 mg: Subjects were administered with MSC2156119J 300 mg once daily for repeated 21-day cycles until disease progression or unacceptable toxicity.
- MSC2156119J 500 mg: Subjects were administered with MSC2156119J 500 mg once daily for repeated 21-day cycles until disease progression or unacceptable toxicity.
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 6
subjects | 0 | 0 | 0

2. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs or TEAEs Leading To Death
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the study drug. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline Up to 30 days after last dose of study drug administration (55.1 weeks)
Population: Safety analysis set included all subjects who had received at least 1 dose of the IMP.
Measure: Number; unit: subjects
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 6
subjects
  TEAEs | 2 | 3 | 6
  Serious TEAEs | 0 | 3 | 1
  TEAEs Leading To Death | 0 | 0 | 1

3. Secondary Outcome: Number of Subjects With Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score of 2 or Higher
Description: ECOG PS score is widely used by doctors and researchers to assess how a subjects' disease is progressing, and is used to assess how the disease affects the daily living abilities of the subject, and determine appropriate treatment and prognosis. The score ranges from Grade 0 to Grade 4, where Grade 0 = Fully active, able to carry on all pre-disease performance without restriction, Grade 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (like light house work, office work), Grade 2 = Ambulatory and capable of all self-care but unable to carry out any work activities, Grade 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours and Grade 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
Time Frame: Baseline up to 30 days after last dose of study drug administration (55.1 weeks)
Population: Safety analysis set included all subjects who had received at least 1 dose of the IMP.
Measure: Number; unit: subjects
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 6
subjects | 0 | 0 | 0

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) After Single Dose of MSC2156119J
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: Pharmacokinetic (PK) analysis set included all subjects who had completed Cycle 1 without any relevant protocol violations with respect to factors that were likely to affect PK results and who received at least first dose of study drug according to protocol providing sufficient concentration time data to determine PK endpoints for the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 6
nanogram per milliliter (ng/mL) | 244.4 (29.9) | 301.3 (42.6) | 442.4 (27.5)

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) After Multiple Dose of MSC2156119J
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: PK analysis set. Here "Number of participants analyzed" signifies those subjects who were evaluable for this outcome at the specified time point for each arm, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 5
ng/mL | 807.5 (11.5) | 610.1 (84.8) | 996.8 (17.5)

6. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) After Single Dose of MSC2156119J
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: PK analysis set included all subjects who had completed Cycle 1 without any relevant protocol violations with respect to factors that were likely to affect the PK results and who received at least first dose of study drug according to the protocol providing sufficient concentration time data to determine the PK endpoints for the study drug.
Measure: Median (Full Range); unit: hours
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 6
hours | 8.000 [7.92 to 8.03] | 8.017 [8.00 to 10.02] | 10.000 [3.97 to 23.85]

7. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) After Multiple Dose of MSC2156119J
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 5
hours | 8.000 [7.98 to 8.02] | 9.917 [1.95 to 10.23] | 4.133 [3.87 to 9.87]

8. Secondary Outcome: Apparent Terminal Half-life (t1/2) of MSC2156119J
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half. Terminal half-life is calculated by dividing the natural logarithm to the base 2 (Ln2) divided by elimination rate constant (λz), where 'λz' is calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1 and Day 14 Cycle 1
Population: It was not possible to calculate data for this outcome measure because dosing interval was too small compared to the long half-life to characterize the terminal phase rate constant, which is needed for the calculation of t1/2.
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Extrapolated Infinite Time (AUC[Inf]) of MSC2156119J
Description: AUC(inf) was calculated by combining AUC0-t and AUCextra. AUCextra represented an extrapolated value obtained by Clast/λz, where Clast was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and λz is the terminal elimination rate constant.
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1 and Day 14 Cycle 1
Population: It was not possible to calculate data for this outcome measure because dosing interval was too small compared to the long half-life to characterize the terminal phase rate constant, which is needed for the calculation of AUCinf.
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Apparent Body Clearance (CL/f) of MSC2156119J
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. CL/F = Dose/AUC(inf), where AUC(inf) =AUC0-t + AUCextra. AUCextra represented an extrapolated value obtained by Clast/λz, where Clast was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and λz is the terminal elimination rate constant.
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1 and Day 14 Cycle 1
Population: It was not possible to calculate data for this outcome measure because dosing interval was too small compared to the long half-life to characterize the terminal phase rate constant, which is needed for the calculation of CL/f.
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Apparent Volume of Distribution Associated To The Terminal Phase (Vz/f) of MSC2156119J
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed and is calculated by Dose/(AUC(inf)*λz).
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1 and Day 14 Cycle 1
Population: It was not possible to calculate data for this outcome measure because dosing interval was too small compared to the long half-life to characterize the terminal phase rate constant, which is needed for the calculation of the Vz/f.
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Sampling Time t (AUC0-t) After Single Dose of MSC2156119J
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration is at or above the lower limit of quantification (LLQ) AUC0-t was calculated according to the mixed log-linear trapezoidal rule
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 1 Cycle 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 6
h*ng/mL | 4060.8 (30.7) | 5412.7 (45.0) | 8235.0 (30.9)

13. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Sampling Time t (AUC0-t) After Multiple Dose of MSC2156119J
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration is at or above the LLQ. AUC0-t was calculated according to the mixed log-linear trapezoidal rule
Time Frame: pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10, 24 hours post-dose on Day 14 Cycle 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- MSC2156119J 200 mg: Subjects were administered with MSC2156119J 215 mg orally once daily for repeated 21-day cycles until disease progression or unacceptable toxicity.
Arm/Group | MSC2156119J 200 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 5
h*ng/mL | 16088.6 (12.2) | 13313.4 (82.5) | 21509.0 (16.7)

14. Secondary Outcome: Number of Subjects With Best Overall Response (BOR)
Description: Number of subjects with BOR in each category (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD]) according to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) was reported. CR: defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: defined as at least a 30% decrease in sum of longest diameter of target lesions, taking as reference the baseline sum of longest diameter. PD: defined as at least a 20% increase in sum of longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or unequivocal progression of existing non-target lesions. SD: defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of longest diameter while on study.
Time Frame: Day 21 of Cycle 2 and each subsequent cycle up to a maximum of 51.1 weeks
Population: Safety analysis set included all subjects who had received at least 1 dose of the IMP.
Measure: Number; unit: subjects
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 6
subjects
  CR | 0 | 0 | 0
  PR | 0 | 0 | 0
  SD | 0 | 0 | 2
  PD | 3 | 3 | 3
  Not Evaluable | 0 | 0 | 1

15. Secondary Outcome: Number of Subjects With Clinical Benefit
Description: Clinical Benefit was defined as CR or PR at any time point or SD at week 12 or later, based on tumor assessment as determined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1). CR: defined as disappearance of all target and all non-target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: defined as at least a 30% decrease in sum of longest diameter of target lesions, taking as reference the baseline sum of longest diameter. SD: defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of longest diameter while on study. PD: defined as at least a 20% increase in sum of longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or unequivocal progression of existing non-target lesions.
Time Frame: Day 21 of Cycle 2 and each subsequent cycle up to a maximum of 51.1 weeks
Population: Safety analysis set included all subjects who had received at least 1 dose of the IMP.
Measure: Number; unit: subjects
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Number analyzed (Participants) | 3 | 3 | 6
subjects | 0 | 0 | 2

16. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time in months from the first administration of trial treatment until first observation of progressive disease (PD), or death due to any cause when death occurs within 12 weeks of the last tumor assessment or first administration of trial treatment (whichever is later). Any subject with neither assessment of tumor progression, nor death within 12 weeks after last tumor assessment date was censored on the date of last tumor assessment. PFS was planned to be presented for "MSC2156119J Combined" reporting arm.
Time Frame: Day 21 of Cycle 2 and each subsequent cycle up to a maximum of 51.1 weeks
Population: Safety analysis set included all subjects who had received at least 1 dose of the IMP.
Measure: Median (90% Confidence Interval); unit: months
Groups:
- MSC2156119J Combined: All subjects who were administered with MSC2156119J 215 mg, 300mg or 500 mg orally once daily for repeated 21-day cycles until disease progression or unacceptable toxicity.
Arm/Group | MSC2156119J Combined
Number analyzed (Participants) | 12
months | 1.38 [1.15 to 1.38]

ADVERSE EVENTS:
Time Frame: Baseline Up to 30 days after last dose of study drug administration (55.1 weeks)
Arm/Group | MSC2156119J 215 mg | MSC2156119J 300 mg | MSC2156119J 500 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/3 | 1/6
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSC2156119J 215 mg (N=3) | MSC2156119J 300 mg (N=3) | MSC2156119J 500 mg (N=6)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
MALAISE (General disorders) | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 0
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MSC2156119J 215 mg (N=3) | MSC2156119J 300 mg (N=3) | MSC2156119J 500 mg (N=6)
FATIGUE (General disorders) | 1 | 2 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 4
MALAISE (General disorders) | 0 | 1 | 1
PYREXIA (General disorders) | 0 | 0 | 1
VESSEL PUNCTURE SITE ERYTHEMA (General disorders) | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 2 | 3
NAUSEA (Gastrointestinal disorders) | 0 | 2 | 3
VOMITING (Gastrointestinal disorders) | 0 | 1 | 3
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 1
ASCITES (Gastrointestinal disorders) | 0 | 1 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 1
PROCTALGIA (Gastrointestinal disorders) | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1 | 3
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 4
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
AMYLASE INCREASED (Investigations) | 0 | 0 | 2
LIPASE INCREASED (Investigations) | 0 | 0 | 2
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 0 | 1
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
TUMOUR ASSOCIATED FEVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
DYSGEUSIA (Nervous system disorders) | 1 | 1 | 1
DIZZINESS (Nervous system disorders) | 0 | 1 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 2
ANXIETY (Psychiatric disorders) | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 1
EYE MOVEMENT DISORDER (Eye disorders) | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 0 | 1
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0
THROMBOPHLEBITIS (Vascular disorders) | 0 | 1 | 0
VARICOSE VEIN (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No